CLINICAL TRIAL: NCT02729623
Title: The Pharmacokinetics, Safety, and Ease of Use of a Portable Metered-Dose Cannabis Inhaler: A Phase 1a Study
Brief Title: The Pharmacokinetics, Safety, and Ease of Use of a Portable Metered-Dose Cannabis Inhaler
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kite Systems (Industry)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cannaHALER-1A
Record Dates: First submitted 2016-03-27; First posted 2016-04-06 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single CannaHALER dose 10 ± 0.1 mg (Experimental): Single dose 10 ± 0.1 mg of cannabis using the Kite Systems CannaHALER cannabis Inhaler device.
  Interventions: Drug: Kite Systems cannaHALER cannabis Inhaler.
- Single CannaHALER dose 15 ± 0.1 mg (Experimental): Single dose 15 ± 0.1 mg of cannabis using the Kite Systems CannaHALER cannabis Inhaler device.
  Interventions: Drug: Kite Systems cannaHALER cannabis Inhaler.
- Single CannaHALER dose 20 ± 0.1 mg (Experimental): Single dose 20 ± 0.1 mg of cannabis using the Kite Systems CannaHALER cannabis Inhaler device.
  Interventions: Drug: Kite Systems cannaHALER cannabis Inhaler.
- Single CannaHALER dose 25 ± 0.1 mg (Experimental): Single dose 25 ± 0.1 mg of cannabis using the Kite Systems CannaHALER cannabis Inhaler device.
  Interventions: Drug: Kite Systems cannaHALER cannabis Inhaler.

INTERVENTIONS:
Drug: Kite Systems cannaHALER cannabis Inhaler.

SUMMARY:
Growing evidence supports the use of inhaled cannabis for neuropathic pain; the lack of standard inhaled dosing holds a major obstacle in cannabis becoming a pharmacological treatment for neuropathic pain. The objective of this study is to explore the pharmacokinetics, safety, tolerability, and ease of use of a portable metered-dose inhaler, (i.e. CannaHALER) for cannabis in a cohort of 12 healthy volunteers. In a single escalating dose methodology, open-label study, patients will inhale a single 10 ± 0.1 mg / 15 ± 0.1 mg / 20 ± 0.1 mg / 25 ± 0.1 mg dose of cannabis using the Kite Systems cannaHALER cannabis Inhaler device. Blood samples will be taken at baseline and up to 30 minutes. Adverse events will be monitored following the inhalation.

ELIGIBILITY:
Inclusion Criteria:

* aged 30-70 years;
* healthy
* if applicable, negative pregnancy test (β human chorionic gonadotropin pregnancy test).

Exclusion Criteria:

* significant cardiac or pulmonary disease,
* history of a psychotic or anxiety disorder,
* pregnancy, pregnancy attempt or breastfeeding,
* presence of a neuropathic or non-neuropathic pain,
* low blood pressure, below 90 mm Hg (systolic)
* Diabetes is diagnosed,
* first degree family history of psychotic or anxiety disorder,
* history of drug addiction,
* history of drug misuse,
* using the following drugs: Rifampicin, Rifabutin, Carbamazepine, Phenobarbital, Primidone,
* using the following plants: Hypericum perforatum, troglitazone,
* Alcohol consumption up to 12 hours before the study,
* abnormal parameters such as Heart Rate above 100 BPM, Blood pressure, below 90 mm Hg (systolic), Saturation below 91 percent,
* Cannabis use up to 12 hours before the study,
* health condition which could affect or alter the experiment results,
* Volunteer has a legal guardian.
* Chronic use of drugs,
* age less than 30 or more than 70,
* a health condition that could affect the outcome of the trial or constitutes a risk factor for participation in the trial.
* The experiment will not include special populations such as pregnant women, children and without judgement.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Δ9-tetrahydrocannabinol levels (THC) | 30 Minutes
Adverse event monitoring | 4 hours
Δ9 Carboxy-THC levels | 30 Minutes

SECONDARY OUTCOMES:
Short Blessed cognitive Test | 30 Minutes
Blood pressure | 120 Minutes
Pulse rate | 120 Minutes
Oxygen saturation | 120 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Ben-Ishay, MD., Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Undecided